CLINICAL TRIAL: NCT03688568
Title: Phase 2 Study of Imatinib in Children With Neurofibromatosis and Airway Tumors
Brief Title: Study of Imatinib in Children With Neurofibromatosis and Airway Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment not feasible
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kent A Robertson, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1505569560; 1R01FD004830-01A2 (FDA)
Record Dates: First submitted 2018-09-11; First posted 2018-09-28 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Neurofibroma, Plexiform
MeSH Terms: conditions — Neurofibroma, Plexiform | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib Mesylate Arm (Experimental): Imatinib Mesylate, given daily orally, 55 mg PO BID, if tolerated for 2 weeks increase to 110 mg/m2 BID, and further increase to 165 and final dosage to 220 mg/m2 bid if tolerated. Can continue for 12 months.
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Imatinib given orally as dose escalation treatment.

SUMMARY:
The purpose of this study is to look at a subset of plexiform neurofibromas and determine if the airway tumors are more sensitive to imatinib therapy. Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged: > 6 months and < 12 years of age.
2. Diagnosis of neurofibromatosis type 1 (NF1).
3. Presence of symptomatic airway plexiform neurofibromas ; defined by abnormal sleep study or pulmonary function testing.
4. Patients must have measurable (> 1.5 cm in two dimensions or able to assess a minimum of 3 slices) disease by magnetic resonance imaging (MRI).
5. Patients must have a Karnofsky of > 70% or Lansky of > 50% and a life expectancy of > 2 months.
6. Adequate end organ function, defined as the following:

   total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L.
7. Patients must be able to swallow whole pills or crushed pills in a soft food such as pudding or apple sauce; or have other GI access such as a G-tube.
8. Written, voluntary informed consent/assent.

Exclusion Criteria:

1. Patient has received any other investigational agents within 14 days of first day of study drug dosing.
2. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
3. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
5. Patient has a known brain metastasis. Non-specific CNS changes on MRI/CT characteristic of NF1 are allowed, but not known CNS malignancies requiring therapeutic intervention.
6. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
7. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
8. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry.
9. Patient previously received radiotherapy to > 25 % of the bone marrow
10. Patient had a major surgery within 2 weeks prior to study entry.
11. Patient/parent with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
12. Patients who have or anticipate receiving permanent (or semi-permanent) metallic structures attached to their body. (e.g., braces on teeth, body piercings), which their physicians believe will interfere with the MRI.
13. Patient has an unstable airway requiring more urgent intervention or deemed unable to travel due to unstable airway by referring MD.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Functional Airway Response | 12 months
  Sleep study or pulmonary function test

SECONDARY OUTCOMES:
Radiologic response of tumor | 12 months
  Volumetric MRI measurements
Quality of Life Assessment | 12 months
  Quality of Life Questionnaire
Cytokine Biomarker | 12 months
  Immunoassay
Inflammatory Cell Biomarker | 12 months
  Flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children - Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No